CLINICAL TRIAL: NCT00700492
Title: Luteal Support With Vaginal Progesterone Capsules Following Ovulation Induction With Human Menopausal Gonadotropins (hMG) for Intra Uterine Insemination: A Comparative Study
Brief Title: Does Hormonal Luteal Support After Intra-uterine Insemination (IUI) Increase the Pregnancy Rate?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in Belgian law on the use of hMG in IUI
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Thomas D'Hooghe, Prof PhD MD, University Hospital, Gasthuisberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML2437-30/12/2003
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Subfertility
Keywords: subfertility; pregnancy rate; miscarriage
MeSH Terms: conditions — Infertility; Abortion, Spontaneous | interventions — Progesterone; Utrogestan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention)
- utrogestan (Experimental): daily use of vaginal progesterone capsules
  Interventions: Drug: progesterone

INTERVENTIONS:
Drug: progesterone — vaginal capsules 3X200mg daily
  Other Names: Utrogestan
  Arms: utrogestan

SUMMARY:
A randomized study to investigate if hormonal luteal support after intra-uterine insemination (IUI) in ovulation induction cycles with human menopausal gonadotropin increases the pregnancy rate

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Tubal patency demonstrated
* ovulation induction with human menopausal gonadotropin

Exclusion Criteria:

* ovulation induction with clomiphene citrate

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2004-05; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate per cycle | 12 weeks pregnancy

SECONDARY OUTCOMES:
rate of miscarriages per cycle | 12 weeks pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Thomad D'Hooghe, MD, PhD, Principal Investigator — University Hospital Gasthuisberg, Catholic University Leuven, Belgium
Locations (1):
- Leuven University Fertility Center, Leuven, Vlaams Brabant, Belgium